CLINICAL TRIAL: NCT06756620
Title: Investigation of the Etiology of Hypertension and Endothelial Damage in Patients With Cytochrome P450 Oxidoreductase Deficiency
Acronym: PORENDO
Status: Completed | Type: Observational
Sponsor: Ozge Bayrak Demirel (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Istanbul University (Other)
Responsible Party: Sponsor-Investigator, Ozge Bayrak Demirel, MD, Istanbul University
Organization: Istanbul University (Other)
Other Study IDs: PORENDO; 324S091 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Cytochrome P450 Oxidoreductase Deficiency; Hypertension; Endothelial Dysfunction; Congenital Adrenal Hyperplasia
Keywords: Cytochrome P450 Oxidoreductase Deficiency; POR Deficiency; Hypertension; Endothelial Dysfunction; Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Antley-Bixler Syndrome Phenotype; Hypertension; Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Venous blood samples will be retained to analyze endothelial damage biomarkers, including Prostaglandin E2, Thromboxane B2, and Nitric Oxide. Serum samples will be centrifuged and stored at -80°C for future biochemical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- POR deficiency: This group includes 7 pediatric patients with genetically confirmed Cytochrome P450 Oxidoreductase (POR) deficiency under follow-up at Istanbul University, Istanbul Faculty of Medicine. The participants will undergo ambulatory blood pressure monitoring (ABPM), nailfold capillaroscopy, and blood sampling for analysis of endothelial damage biomarkers (Prostaglandin E2, Thromboxane B2, and Nitric Oxide). These patients are currently receiving physiologic doses of hydrocortisone as part of their standard care.
- Healthy Control Group: This group consists of 30 healthy children and adolescents recruited from Istanbul University, Istanbul Faculty of Medicine. Participants are age- and gender-matched to the POR deficiency group. They will undergo ambulatory blood pressure monitoring (ABPM), nailfold capillaroscopy, and blood sampling for analysis of endothelial damage biomarkers (Prostaglandin E2, Thromboxane B2, and Nitric Oxide). These participants have no known medical conditions or history of chronic illness.

SUMMARY:
This study investigates the etiology of hypertension and endothelial damage in patients with Cytochrome P450 Oxidoreductase (POR) deficiency. The study involves comparing ambulatory blood pressure monitoring (ABPM), endothelial biomarkers (Prostaglandin E2, Thromboxane B2, and Nitric Oxide levels), and capillaroscopy findings between POR deficiency patients and healthy controls.

DETAILED DESCRIPTION:
Cytochrome P450 Oxidoreductase (POR) deficiency is a rare autosomal recessive condition associated with congenital adrenal hyperplasia and other systemic complications. This study aims to elucidate the role of endothelial dysfunction and hypertension in POR deficiency by comparing the biochemical, vascular, and clinical parameters of POR-deficient patients with age- and gender-matched healthy controls. The research could pave the way for targeted therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of Cytochrome P450 Oxidoreductase (POR) deficiency
* Diagnosis of POR deficiency before the age of 18.
* Written informed consent provided by the participant and/or their legal guardian.

Exclusion Criteria:

* Presence of an acute illness or other pathology identified during the study. Nail-biting habit or manicure within the last 14 days (due to potential impact on capillaroscopy results)
* Use of medications other than physiologic hydrocortisone
* Kidney, endocrine, or vascular pathologies that may cause hypertension
* History of smoking or hand trauma

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of two groups: (1) 7 pediatric patients with genetically confirmed Cytochrome P450 Oxidoreductase (POR) deficiency under follow-up at Istanbul University and (2) 30 healthy children and adolescents matched by age and gender, without any known medical conditions. The population aims to evaluate the impact of POR deficiency on hypertension and endothelial damage.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Serum Endothelial Biomarkers (Prostaglandin E2, Thromboxane B2, and Nitric Oxide) in POR Deficiency Patients Compared to Healthy Controls | Up to 6 months from the start of participant enrollment
  This measure evaluates the serum levels of endothelial biomarkers, including Prostaglandin E2, Thromboxane B2, and Nitric Oxide, to determine differences between patients with Cytochrome P450 Oxidoreductase (POR) deficiency and healthy controls. These biomarkers are critical for assessing endothelial dysfunction, which may contribute to hypertension in POR deficiency patients.

SECONDARY OUTCOMES:
Ambulatory Blood Pressure Monitoring (ABPM) Findings in POR Deficiency Patients Compared to Healthy Controls | Up to 6 months from the start of participant enrollment
  This measure assesses the 24-hour ambulatory blood pressure monitoring (ABPM) results, including systolic, diastolic, and mean arterial pressures, in Cytochrome P450 Oxidoreductase (POR) deficiency patients compared to healthy controls. It aims to identify hypertension prevalence and nocturnal blood pressure patterns in POR deficiency patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Bayrak Demirel, MD, Study Director — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will not be shared due to confidentiality concerns and the small sample size of the study, which may risk participant anonymity.